CLINICAL TRIAL: NCT01934907
Title: Transfusion Reaction by Washed Red Blood Cell (RBC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-1307/212-009
Record Dates: First submitted 2013-08-22; First posted 2013-09-04 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- washed RBC (Experimental): Packed RBCs are Washed and then, transfused.
  Interventions: Other: Washing of packed RBC by normal saline
- pack RBC (No Intervention): Packed RBCs are transfused.

INTERVENTIONS:
Other: Washing of packed RBC by normal saline
  Arms: washed RBC

SUMMARY:
The hypothesis is that transfusion of washed red blood cell can decrease the complication by transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total hip replacement arthroplasty

Exclusion Criteria:

* Patients who do not agree with this clinical study.
* Patients who have a history of transfusion for recent 1 month.
* Patients who have rare blood types.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Complication by transfusion | Operation day and during postoperative 5 days

SECONDARY OUTCOMES:
Total units of RBC transfused. | On the operation day and during the postoperative 5 days
Hemoglobin | 1 day before the operation day and postoperative 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea